CLINICAL TRIAL: NCT06439446
Title: The Effect of Family Characteristics on the Functional Level of Children With Cerebral Palsy of the Spastic Type With Walking Ability
Brief Title: Functionality and Family Characteristics in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Atahan TURHAN, Principal Investigator, Dr. Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: KAEU-T.ATAHAN-004
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Family Characteristics
Keywords: Functional Level
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to investigate the effect of family characteristics on functional level in children with Spastic Type Cerebral Palsy who are able to walk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hemiparetic and diparetic type CP
* Between the ages of 5-15
* GMFCS level I, II and III
* Volunteer individuals were included.

Exclusion Criteria:

* Having undergone a surgical operation within the last year,
* Having contracture in the lower extremity,
* Having had a fracture in the lower extremity in the last 6 months,
* Botulinum Toxin A (BTX-A) administered in the last 6 months
* Patients with cognitive, visual or hearing impairments that would prevent communication with their peers and siblings were excluded from the study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study was carried out at Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center. Patients who applied to the Physical Medicine and Rehabilitation Polyclinic with the diagnosis of CP were examined by a physical therapist. Parents of children who met the inclusion criteria were interviewed and informed about the study.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Level | 36 week
  Gross motor function level was measured with Gross Motor Function Measure-66 (GMFM-66). GMFM-66 is a 66-item test developed to measure gross motor skills in children with cerebral palsy and can be evaluated in 5 different categories, including reaching and rolling, sitting, crawling and crawling, standing, walking, running and jumping. It is a 4-point Likert type scale. Higher scores on the test indicate higher gross motor skills.
Parents' Quality of Life | 36 week
  Parents' self-reported quality of life functions such as physical, emotional, social, and cognitive were assessed with The PedsQL Family Impact Module. Total score range is 0-100. Higher scores on the scale indicate less anxiety.

SECONDARY OUTCOMES:
Gross Motor Function Classification | 36 week
  Gross motor functional classification was evaluated with the Gross Motor Function Classification System (GMFCS). GMFCS classifies children with Cerebral Palsy into 5 levels (1-5) based on their motor skills, functional abilities, assistive technologies, and wheelchair needs.
Sociodemographic Form | 36 week
  Characteristic information about the family, such as the family's average monthly income, the number of people living in the family, and the region in which the family lived, was collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turhan A, Kurt-Aydin M, Tarsuslu T. Determinants of Gross Motor Function in Children With Ambulatory Spastic Cerebral Palsy: A Cross-Sectional Study in Turkey. J Paediatr Child Health. 2025 May;61(5):795-801. doi: 10.1111/jpc.70034. Epub 2025 Mar 18. PMID 40099358